CLINICAL TRIAL: NCT02705261
Title: Coaching for Confidence: Evaluating an Internet-based Program to Help Parents Help Children With Difficulty With Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. John Walker, Professor, Dept of Clinical Health Psychology, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 246529
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Anxiety Disorders
Keywords: child; behavior therapy; cognitive therapy; parent; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive-behavior therapy (Experimental): Cognitive-behavior therapy to teach parents the skills to help their children. Participants will have access to the program as often as they wish and have the post assessment at week 12.
  Interventions: Behavioral: cognitive-behavior therapy

INTERVENTIONS:
Behavioral: cognitive-behavior therapy — Internet based program to support parents in developing strategies to help their children

SUMMARY:
The study is an open trial to evaluate a web-based intervention. The intervention focuses on supporting parents to help their children to overcome problems with anxiety. The children who are the focus of the study are in the age ranges of 4 - 12 and experience problems with separation anxiety, social anxiety, or generalized anxiety as identified by their parents. The program will exclude obsessive-compulsive disorder and post-traumatic stress disorder that are seen less often in this age group and require somewhat different interventions.

DETAILED DESCRIPTION:
Parents will be recruited for the study through stories in the media and notices sent through the schools to parents of school age children. The information will invite parents to contact the study staff if in their view their child is more anxious, fearful, shy or worried than most children of their age. Parents will be screened to insure that the child's problem is appropriate for the study. If the child and family are judged to be appropriate for the study they will be provided a user name and password to access a web-based program called Coaching for Confidence. In the first part of the program they review the consent form and decide if they wish to provide consent. If they provide consent they complete initial assessment measures describing their child and themselves. Once the assessment is completed they have access to the program through the internet. They are encouraged to complete the program over a period of 10 weeks. The program focuses on supporting the parent's understanding of child anxiety and the strategies they can take in helping their child to overcome limitations related to anxiety.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of social anxiety, separation anxiety, or generalized anxiety disorder
* judged by parent to have anxiety that interferes with functioning in the home or school.
* judged by clinician to have anxiety that interferes with functioning in the home or school.
* parent unable to read and write in English.
* parent unable to access the internet regularly - at least once a week

Exclusion Criteria:

* diagnosis of obsessive compulsive disorder
* diagnosis of post-traumatic stress disorder
* diagnosis of school refusal and not attending school at least half of the time
* diagnosis of selective mutism
* diagnosis of autism spectrum disorder
* diagnosis of pervasive developmental disorder
* child currently receiving psychosocial treatment for anxiety

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Spence Children's Anxiety Scale - Parent-rated | 12 weeks
  Rating scale describing a child's anxiety symptoms - 39 items

SECONDARY OUTCOMES:
Clinical Global Improvement Scale - parent confidence | 12 weeks
  7 point rating scale indicating parent confidence in helping child with anxiety
Clinical Global Improvement Scale - child anxiety | 12 weeks
  7 point rating scale indicating degree of improvement or worsening in child anxiety

CONTACTS AND LOCATIONS:
Overall Officials: John R. Walker, Ph.D., Principal Investigator — University of Manitoba, College of Medicine
Locations (1):
- University of Manitoba, College of Medicine, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No